CLINICAL TRIAL: NCT06529562
Title: Surgery Plus Reduced Target Chemoradiotherapy Versus Surgery Plus Reduced Dose Chemoradiotherapy for Newly Diagnosed Operable Nasopharyngeal Carcinoma : a Prospective, Multicenter, Radomized Control Trial
Brief Title: Surgery Plus Reduced Target Chemoradiotherapy vs Surgery Plus Reduced Dose Chemoradiotherapy for Newly Diagnosed Operable Nasopharyngeal Carcinoma.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ming-Yuan Chen (Other)
Collaborators: Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-sen University (Other); Fifth Affiliated Hospital of Guangzhou Medical University (Other); Huazhong University of Science and Technology Union Hospital (Nanshan Hospital) (Unknown); The First Affiliated Hospital of University of South China (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Nanchang City First Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Ming-Yuan Chen, Professior, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-20240221
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Surgery; Target-Reduction Chemoradiotherapy; Dose-Reduction Chemoradiotherapy; Locally Resectable Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery plus target reduction Chemoradiotherapy (Active Comparator): Surgery:
  Endoscopic Nasopharyngectomy:Radical Reaction of the Primary Lesion Using Nasal Endoscopy.
  Retropharyngeal lymphadenectomy: Radical retropharyngeal LNs reaction using nasal endoscopy.
  Neck lymph node dissection Selection of region where the possitive lymph nodes are located.
  Intensity modulated radiotherapy with GTV and CTV1 Reduction:
  CTV2:50.00Gy/25Fr/2.00Gy. Chemotherapy: cisplatin-based regimens.
  Interventions: Radiation: Surgery combined with Target-reduction intensity-modulated radiotherapy
- surgery plus dose reduction Chemoradiotherapy (Experimental): Surgery:
  Endoscopic Nasopharyngectomy: Radical Reaction of the Primary Lesion Using Nasal Endoscopy.
  Retropharyngeal lymphadenectomy: Radical retropharyngeal LNs reaction using nasal endoscopy.
  Neck lymph node dissection Selection of region where the possitive lymph nodes are located.
  Intensity modulated radiotherapy with CTV1 and CTV2 dose Reduction:
  CTV1：48.00-50.00Gy/20Fr/2.40-2.50Gy； CTV2：40.00Gy/20Fr/2.00Gy. Chemotherapy: cisplatin-based regimens.
  Interventions: Radiation: Surgery combined with Dose-reduction intensity-modulated radiotherapy

INTERVENTIONS:
Radiation: Surgery combined with Target-reduction intensity-modulated radiotherapy — in control arm
  Other Names: Target-reduction intensity-modulated radiotherapy
  Arms: surgery plus target reduction Chemoradiotherapy
Radiation: Surgery combined with Dose-reduction intensity-modulated radiotherapy — in experimental arm
  Other Names: Dose-reduction intensity-modulated radiotherapy
  Arms: surgery plus dose reduction Chemoradiotherapy

SUMMARY:
The goal of this clinical trial is to compare surgery plus reduced target chemoradiotherapy with surgery plus reduced dose chemoradiotherapy in newly diagnosed operable Nasopharyngeal Carcinoma.The main questions it aims to answer are:whether endoscopic surgery combined with reduced dose chemoradiotherapy vs surgery plus target reduction chemoradiotherapy can bring substantial survival benefits, lower toxicity, and shorter treatment cycle for patients with operable nasopharyngeal carcinoma .

DETAILED DESCRIPTION:
Currently, the treatment of newly diagnosed non-metastatic nasopharyngeal carcinoma with intensity modulated radiotherapy as the core and chemotherapy with platinum-containing drugs has achieved good therapeutic outcomes. However, the toxicity and side effects caused by local radiotherapy greatly affect the quality of life of patients with nasopharyngeal carcinoma during treatment. In order to find a more "high-efficiency and low-toxicity" nasopharyngeal cancer treatment mode, combined with minimally invasive surgery for radical tumor treatment and radiotherapy and chemotherapy to eliminate potential micro-metastatic lesions,, Our team has previously carried out "prospective clinical trial of newly diagnosed operable nasopharyngeal carcinoma surgery combined with reduced target chemoradiotherapy versus conventional chemoradiotherapy", It has been prelim natively confirmed that gross tumor volume(GTV) and clinical tumor volume (CTV1) high-risk infiltrating area need not be recharacterized after the combined nasopharyngeal or non-combined retropharyngeal surgery and radical resection of cervical lesions. Only low risk infiltrating area (CTV2) was delineated and preventive irradiation of 54 Gy/33 times /45 days was administered, combined with induction or concurrent chemotherapy. Preliminary study results showed that it could further reduce the local recurrence of tumors and the overall curative effect while reducing the toxic side effects of treatment and achieve the therapeutic effect of increased efficacy and reduced toxicity.

Although compared to the conventional radiotherapy dose of 70Gy, postoperative reduced target radiotherapy has achieved a significant reduction in radiotherapy dose while ensuring tumor control, However, we are concerned that nearly 40% of patients still have ≥ grade 3 dry mouth, mucosal ulcer, mouth difficulty and dysphagia during or after treatment. Therefore, for newly diagnosed patients with surgically resectable nasopharyngeal carcinoma, we plan to conduct a prospective clinical trial comparing the survival prognosis and toxic side effects of newly diagnosed surgery combined with reduced dose radiotherapy compared with conventional reduced target radiotherapy combined with concurrent chemotherapy. To explore whether this treatment model can bring comparable survival benefits, lower toxic side effects and shorter treatment cycles for patients.

According to our team's previous research results and literature data, we designed the following scheme: patients with operable nasopharyngeal carcinoma were assigned to the control group and the experimental group. Control group: nasopharyngeal combined with or without combined retropharyngeal and neck lesions radical surgery, postoperative routine target reduction chemoradiotherapy at the same period. Experimental group: Patients underwent radical surgery with or without nasopharynx combined with retropharyngeal and cervical lesions, followed by concurrent low-dose radiotherapy and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Performance Status Score 0-1 points.
* Non-keratinized carcinoma of the nasopharynx (differentiated or undifferentiated, i.e., WHO type II or III) confirmed histologically and/or cytologically.
* Patients with primary nasopharyngeal lesions evaluated as surgically resectable, including T1 (tumor limited to nasopharynx), T2 (tumor limited to the surface of parapharyngeal space) and T3 (tumor limited to the bottom wall of sphenoid sinus) and tumor diameter ≤1.5cm. Resectable retropharyngeal lymph nodes were defined as; The diameter was ≤ 1.5cm, the tissue space was intact, and there was no obvious extranodal invasion; The resectable cervical lymph nodes were defined as ≤ 3cm in diameter, located above the lower edge of the cricoid cartilage, with moderate mobility and no obvious extranodal invasion. Clinical stage: T1-3N1-2M0, T2-3N0M0 (Stage II-III) according to AJCC 8th staging edition.
* Adequate organ function: WBC ≥ 4×10^9 /L, NEUT ≥ 2×10^6 /L, HGB ≥ 9 g/dL, PLT count ≥ 100×10^9/L, TBIL ≤1.5 ULN (TBIL ≤3 ULN for patients with Gilbert Disease), ALT ≤3 ULN, AST ≤3 ULN, ALP ≤3 ULN, ALB ≥ 3 g/dL, INR or APTT≤1.5 ULN, Scr ≤1.5 ULN or Ccr ≥ 60 mL/min.
* Informed Concent signed with willingness to obey the follow-up, treatment, examination and any other programs according to the research protocol.

Exclusion Criteria:

* Diagnosed as recurrent or distant metastatic nasopharyngeal carcinoma or together with any other malignancy.
* Suffering severe organ dysfunction or physical disorder which could not tolerate surgery or radiotherapy or chemotherapy.
* Retropharyngeal lymph node diameter>1.5cm, or extranodal invasion, such as invasion of internal carotid artery, muscle, or extensive extracapsular dissemination.
* Cervical lymph node diameter>3cm, or in the area below the lower margin of the cricoid cartilage, or with extranodal invasion, such as invasion of the internal carotid artery, skin, muscle, mediastinal structure, prevertebral fascia or cervical spine, or extensive extra-capsular spread, subcutaneous metastasis, etc.
* Unable to cooperate with regular follow-up due to psychological, social, domestic or geological reasons.
* During pregnancy or lactation.
* Other patients that the chief physician considered as illegal for this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2032-11-01 (Estimated); Study Completion 2032-11-01 (Estimated)

PRIMARY OUTCOMES:
Locoregional Recurrence-Free Survival Time (LRRFS) | 3 years
  The time interval between randomization and locoregional recurrence, or censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  The OS was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.
Incidence of Treatment-Related Adverse Events | 1 years
  The proportion of patients with treatment related adverse events according to NCI-CTCAE 5.0 and RTOG criteria.
Distant Metastasis-Free Survival (DMFS) | 3 years
  The DMFS is evaluated and calculated from the date of random assignment until the day of first distant metastases or censored at the date of the last follow-up.
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) before treatment, during treatment, after treatment and follow up.
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) | 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) before treatment, during treatment, after treatment and follow up.
Progression-Free Survival (PFS) | 3 years
  The PFS was defined as the duration from the date of random assignment to the date of disease progression or censored at the date of the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD,PhD, Principal Investigator — SUN yet-sen University
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China